CLINICAL TRIAL: NCT07381608
Title: Clinical and Patient-reported Outcomes of Guided Versus Freehand Harvesting Of Positioning of Autogenous Bone Shells: a Randomized Controlled Trial
Brief Title: Clinical and Patient-reported Outcomes of Guided Versus Freehand Harvesting Of Positioning of Autogenous Bone Shells
Acronym: guided
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shalash Dental education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 25-055
Record Dates: First submitted 2026-01-17; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Alveolar Bone Loss in Mandible; Guided Bone Regeneration; Dental Implant
Keywords: alveolar ridge augmentation; guided bone regeneration; dental implant

STUDY DESIGN:
Intervention Model Description: Two arm parallel randomized controlled clinical trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Free hand (Active Comparator): Participants in this arm will undergo vertical ridge augmentation using the conventional freehand shell technique. Thin cortical bone plates will be harvested manually from the donor site and positioned at the recipient site without guides, relying on surgeon experience and judgment. The shells will be fixed with microscrews, filled with autogenous bone chips, and covered with a resorbable collagen membrane before suturing. This represents the current standard method of care.
  Interventions: Device: Free hand shell technique
- Guided shell technique (Experimental): Participants in this arm will undergo vertical ridge augmentation using the conventional freehand shell technique. Thin cortical bone plates will be harvested manually from the donor site and positioned at the recipient site without guides, relying on surgeon experience and judgment. The shells will be fixed with microscrews, filled with autogenous bone chips, and covered with a resorbable collagen membrane before suturing. This represents the current standard method of care.
  Interventions: Device: Guided shell technique

INTERVENTIONS:
Device: Free hand shell technique — In this group, a 3D scan of the patient's jaws will be taken. Using specialized computer software, the surgeon will design custom guides for harvesting the bone shell and positioning it at the recipient site. These guides are then 3D-printed. During surgery, the guides fit onto the patient's jaw and direct the cutting and placement of the bone shell with high precision. This process is expected to shorten the procedure and reduce errors.
  Arms: Free hand
Device: Guided shell technique — Participants in this arm will undergo vertical ridge augmentation using the conventional freehand shell technique. Thin cortical bone plates will be harvested manually from the donor site and positioned at the recipient site without guides, relying on surgeon experience and judgment. The shells will be fixed with microscrews, filled with autogenous bone chips, and covered with a resorbable collagen membrane before suturing. This represents the current standard method of care.
  Arms: Guided shell technique

SUMMARY:
When people lose teeth or have gum disease, the jawbone can shrink over time. This shrinkage makes it difficult for dentists to place dental implants because implants need a strong and stable base of bone. To solve this problem, surgeons often use bone grafting techniques. One of the most reliable ways to rebuild lost bone is called the autogenous shell technique. In this method, very thin plates of bone are taken from another part of the patient's mouth, shaped into a "shell," and fixed into place at the site where bone is missing. The empty space inside the shell is then filled with tiny bone chips, and the whole graft heals into strong new bone over time. Once healed, implants can be placed securely.

This technique has been widely studied and is considered highly effective. However, it is not easy to perform. Traditionally, the shells are harvested and positioned by hand, relying heavily on the skill and experience of the surgeon. Even very experienced clinicians face challenges: the shells can break if cut too thin, positioning may take a long time, and results can vary from patient to patient. Patients also report significant discomfort after surgery, including swelling, pain, and difficulty eating and speaking during recovery.

In recent years, digital technology has begun to transform oral surgery. Using 3D imaging and computer design, it is now possible to create custom surgical guides and positioning jigs. These guides are printed with 3D printers and act like templates, helping surgeons cut bone in exactly the right size and shape, and place it precisely in the planned position. In implant dentistry, such guides are already used for the accurate placement of dental implants, and studies show they can make surgery faster and safer. However, little is known about whether these guides also improve patient comfort and recovery when used in bone grafting procedures such as the shell technique.

This clinical trial has been designed to answer that question. It compares two groups of patients who need vertical bone augmentation before implant placement:

Guided group: Patients treated with 3D-printed surgical guides for harvesting and positioning bone shells.

Freehand group: Patients treated with the conventional freehand shell technique without guides.

By studying both groups, the trial aims to determine whether guided surgery reduces pain, swelling, and recovery problems, and whether it saves time in the operating room. Most importantly, it seeks to put patients' voices at the center by focusing on patient-reported outcome measures (PROMs)-direct feedback from patients about how they feel after the procedure.

DETAILED DESCRIPTION:
Why This Trial is Needed. Bone augmentation surgeries are elective procedures. Patients choose them to improve their quality of life through implant-supported teeth. Because these surgeries are optional, patients' comfort, recovery, and satisfaction are especially important. Traditional studies often measure only technical outcomes, such as how much bone is gained or whether implants survive in the long term. While these outcomes are essential, they do not tell the whole story. A patient may have a technically successful bone graft but still feel the experience was very painful or difficult, which could reduce trust in dental care.

The guided shell technique holds promise for reducing patient suffering. By making surgery quicker and more precise, it might limit tissue trauma and shorten healing time. Yet, until now, no high-quality randomized controlled trial (RCT) has compared guided versus freehand shell grafting from the patient's perspective. This lack of evidence is a gap that needs to be filled so that patients and clinicians can make informed choices. If guided surgery proves superior, it could become the new standard of care, ensuring safer and more comfortable treatment for people needing implants.

Purpose of the Study

The main goal of this study is to compare the patient-reported outcomes between guided and freehand autogenous shell grafting. Specifically, the trial will investigate:

How much pain, swelling, bruising, difficulty chewing, and limited mouth opening (trismus) patients experience after surgery.

Whether patients feel more comfortable overall when treated with guides. How many painkiller tablets do patients need during the first week after surgery? How long does the operation take in each group? Whether complications such as infection or graft failure occur more often in one method than the other.

By looking at these factors, the trial will provide a complete picture of not just how well the bone graft works, but how patients actually feel throughout recovery.

Study Design: This research is a prospective randomized controlled clinical trial. That means patients are enrolled before the surgery, randomly assigned to one of two groups, and followed over time to measure outcomes. Randomization is important because it ensures that the two groups are similar at the start, so any differences in results can be attributed to the surgical method rather than patient characteristics.

The study will recruit 54 patients in total. Each patient will be randomly placed into either the guided group (27 patients) or the freehand group (27 patients). This number was carefully calculated based on statistical formulas to ensure the study has enough power to detect meaningful differences, especially in reported pain levels.

The trial will be conducted at the Shalash Dental Centre clinic.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-99years. Classified as American Society of Anesthesiologists (ASA) I or II.
* Partial edentulism (missing teeth) requiring ≥4 mm vertical ridge augmentation.
* Presence of a suitable intraoral donor site for bone harvesting.
* Good oral hygiene, with Full Mouth Plaque Score (FMPS) < 25%.

Exclusion Criteria:

* Systemic contraindications to oral surgery (uncontrolled systemic disease). -History of head or neck radiotherapy.
* Current or past use of bisphosphonates or other medications affecting bone healing.
* Smokers of more than 10 cigarettes per day.
* Pregnant or breastfeeding women.
* Presence of active oral infection at the surgical site.
* Untreated periodontal disease.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain (0-10) | 7 days
  The Visual Analogue Scale for Pain is a Likert scale (0-10) in which the patient rates pain in response to prespecified questions (Pilowsky and Kaufman, 1965). This is a standard tool for recording subjective measurements, such as pain, into a measurable outcome that can be compared across subjects enrolled in the study. On this scale 0 means there is no pain felt, and 10 is the worst possible pain felt. Lower scores indicate lower pain and higher scores indicate severe pain.

SECONDARY OUTCOMES:
analgesic intake | 7 days
  Analgesic intake will be recorded by the patient as the number of tablets and frequency, and will be measured in mg totally after 1 week, the higher the number of mg of analgesic would indicate severe pain and discomfort while low analgesic intake would indicate low pain.
Surgical time | on the day of the surgery ( T1)
  The amount of time for the procedure will be recorded in minutes during the intervention and the control procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud shalash, PhD, Principal Investigator — National Research Centre Cairo Egypt
Locations (1):
- Shalash Implant Education, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No